CLINICAL TRIAL: NCT04510753
Title: Evaluation of Sensifree's Algorithm for Continuous Blood Pressure Measurements Based on a PPG Sensor's Signal Compared to Invasive Radial Arterial Line
Brief Title: Data Collection of Arterial Line Waveform and BP Values
Status: Completed | Type: Observational
Sponsor: Sensifree Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-30-0054
Record Dates: First submitted 2020-07-29; First posted 2020-08-12 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2020-08

CONDITIONS: Blood Pressure Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Arterial catheterization kit — Invasive monitoring of blood pressure via catheterization of the radial artery, displaying a continuous pressure waveform and blood pressure values.
Device: GE Datex-Ohmeda Finger Clip Pulse Oximeter Sensor — PPG fingertip mounted sensor, that measures the oxygen level (oxygen saturation) of the blood and generates a waveform
Device: NIBP Cuff (GE Healthcare) — A blood pressure cuff is used to measure blood pressure. The cuff has an inflatable rubber bladder that is typically fastened around the arm. A pressure meter indicates the cuff's pressure.

SUMMARY:
Collect continuous systolic and diastolic blood pressure values and waveforms as recorded by an arterial line catheter and by non-invasive blood pressure (NIBP) and to collect Photoplethysmogram Pulse Oximetry (PPG) waveform in order to optimize the Sensifree algorithm.

DETAILED DESCRIPTION:
Sensifree is developing a continuous non-invasive blood pressure measurement system, that uses a fingertip PPG sensor as a signal source. The system provides systolic, diastolic and mean arterial pressure values, for use in hospitals and other clinical settings. The PPG waveform is analyzed by a proprietary software algorithm, calculating BP values.

The current best method to obtain similar information is by using an Arterial line catheter which will serve as a reference device. In this study, the sponsor aims to prospectively collect continuous radial arterial line & PPG waveforms, as well as NIBP data over the period of the surgery in order to test and refine the algorithm.

ELIGIBILITY:
Inclusion Criteria:

1. Signed inform consent
2. Age 18 or greater
3. Elective surgery that requires invasive BP monitoring (A-line)

Exclusion Criteria:

1. Emergency surgery
2. A-line not inserted
3. Informed consent not signed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery involving placement of radial artery A-line for BP monitoring
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
Comparison of BP values between a PPG sensor based device and an arterial line | The length of each procedure, typically up to 8 hours
  PPG signal will be acquired from the PPG sensor, while blood pressure values (systolic, diastolic, mean) will be acquired from A-line. PPG signal will be analyzed by the Sensifree's algorithm and compared to the A-line BP measurement results according to ISO 81060-2 accuracy specifications

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Wallace, MD, PhD, Principal Investigator — San Francisco Veterans Affairs Medical Center
Locations (1):
- San Francisco Veterans Affairs Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No